CLINICAL TRIAL: NCT01296451
Title: A Phase I Study to Assess the Safety and Immunogenicity of AdCh3NSmut and MVA-NSmut in Healthy Volunteers and Patients With Hepatitis C Virus Infection
Brief Title: Study of a New MVA Vaccine for Hepatitis C Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReiThera Srl (Industry)
Collaborators: University of Oxford (Other); Oxford University Hospitals NHS Trust (Other); University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV003; 2009-018260-10 (EudraCT Number)
Record Dates: First submitted 2011-02-09; First posted 2011-02-15 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C; vaccine; Adenovirus; MVA; chronic infection; interferon; ribavirin
MeSH Terms: conditions — Hepatitis C; Adenoviridae Infections; Persistent Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Arm A, group1 (Experimental): Intervention: MVA-NSmut. Administration schedule: 1 dose MVA-NSmut 2 x 10^8 pfu. Subjects: 4 healthy volunteers
  Interventions: Biological: MVA-NSmut
- Arm A, group 2 (Experimental): Interventions: AdCh3NSmut; MVA-NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at week 0 and 1 dose MVA-NSmut 2 x 10^8 pfu at week 8.
  Subjects: 10 healthy volunteers
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut
- Arm B, group 1 (Experimental): Interventions: AdCh3NSmut; MVA-NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at week 14 and 1 dose MVA-NSmut 2 x 10^8pfu at week 22, after starting PEG-IFN and ribavirin therapy.
  Subjects: 5 patients
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut
- Arm B, group 2 (Experimental): Interventions: AdCh3NSmut; MVA-NSmut.. Administration schedule: 1 dose AdCh3NSmut 2.5 x 1010vp at week 2 and 1 dose MVA-NSmut 2 x 108pfu at week 10, after starting PEG-IFN and ribavirin therapy.
  Subjects: 5 patients
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut
- Arm C, group 1 (Experimental): Interventions: AdCh3NSmut; MVA-NSmut Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at week 0 and 1 dose MVA-NSmut 2 x 10^8pfu at week 8.
  Subjects: 4 patients
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut
- Arm A, group 3 (Experimental): Interventions: AdCh3NSmut; MVA-NSmut Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp at week 0, 1 dose MVA-NSmut 2 x 10^8pfu at week 8, 1 dose AdCh3NSmut 2.5 x 10^10vp at week 16 and 1 dose MVA-NSmut 2 x 10^8 pfu at week 24.
  Subjects: 5 healthy volunteers
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut
- Arm A, group 4 (Experimental): Intervention: AdCh3NSmut; MVA-NSmut. Administration schedule: 1 dose AdCh3NSmut 2.5 x 10^10vp (at least 6 months after they were initially enrolled) and 1 dose MVA-NSmut 2 x 10^8 pfu 8 weeks later.
  Subjects: up to 5 healthy volunteers who were previously in group A2
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut
- Experimental: Arm A, group5 (Experimental): Intervention: AdCh3NSmut1. MVA-NSmut. Administration schedule:1 dose AdCh3NSmut1 2.5 x 10^10vp at week 0, 1 dose MVA-NSmut 2 x 10^8 pfu at week 8 and 1 dose MVA-NSmut 2 x 10^8 pfu at week 40.
  Subjects: 5 healthy volunteers
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut1
- Arm A, group 6 (Experimental): Interventions: AdCh3NSmut1. Administration schedule: 1 dose AdCh3NSmut1 2.5 x 10^10 vp at week 0 and 1 dose MVA-NSmut 2 x 10^7 pfu at week 8.
  Subjects: 5 healthy volunteers
  Interventions: Biological: AdCh3NSmut1
- Arm A, group 7 (Experimental): Interventions: AdCh3NSmut1; MVA-NSmut. Administration schedule: 1 dose AdCh3NSmut1 2.5 x 10^10 vp at week 0 and 1 dose MVA-NSmut 2 x 10^6 pfu at week 8.
  Subjects: 5 healthy volunteers
  Interventions: Biological: MVA-NSmut; Biological: AdCh3NSmut1

INTERVENTIONS:
Biological: MVA-NSmut — Genetic vaccine against Hepatitis C virus infection
  Arms: Arm A, group 2; Arm A, group 3; Arm A, group 4; Arm A, group 7; Arm A, group1; Arm B, group 1; Arm B, group 2; Arm C, group 1; Experimental: Arm A, group5
Biological: AdCh3NSmut — genetic vaccine against Hepatitis virus infection
  Arms: Arm A, group 2; Arm A, group 3; Arm A, group 4; Arm B, group 1; Arm B, group 2; Arm C, group 1
Biological: AdCh3NSmut1 — genetic vaccine against Hepatitis virus infection
  Arms: Arm A, group 6; Arm A, group 7; Experimental: Arm A, group5

SUMMARY:
The study is aimed at assessing the safety of AdCh3NSmut and the new candidate vaccine MVA-NSmut when administered sequentially, or alone, to healthy volunteers and patients with hepatitis C virus infection The study also aims at assessing the cellular immune response generated by AdCh3NSmut and MVA-NSmut administered as mentioned above.

DETAILED DESCRIPTION:
The scientific rationale supporting this study can be summarised as follows: an effective antiviral T cell response can mediate HCV viral control and induce the spontaneous resolution of HCV during primary infection. This observation strongly supports the case for the development of T cell induction strategies as a potential therapy for HCV. A hallmark of persistent HCV infection, when viral loads are high, is a weak and narrowly focused HCV specific T cell response, whereas in resolved infection with undetectable viral loads robust T cell responses are detected. Furthermore, mouse and other human models of persistent viral infection show that antigen load crucially determines the quality and quantity of the anti-viral T cell responses so generated [17-18]. This supports the case for the assessment of efficacy of T cell induction, a) in the setting of low viral loads following viral suppression with combination therapy, and b) in the setting of high viral loads. Since pre-existing anti-vector immunity to adenoviral vectors may limit vaccine efficacy, we have conducted a phase-I clinical trial in healthy human subjects using human (Ad6) and simian (AdCh3) adenoviral vectors found at low sero-prevalence in human populations, in a heterologous prime/boost regimen (study HCV001). The same vectors are also under investigation in HCV infected patients (HCV002). These vectors encode the HCV non-structural proteins with a genetically inactivated polymerase gene (NSmut). We have shown that both vectors are safe and highly immunogenic. In preclinical primate studies using identical vectors, heterologous boosting increased peak responses and long-term immunity. However, in humans it appears that, although HCV specific T-cell responses increase following boosting, the magnitude of this response is reduced compared to that observed during vaccine priming. This is probably due to the induction of cross-reactive immunity between the two vectors. In contrast, it has recently been shown that Modified Vaccinia Ankara (MVA) encoding the malaria antigen ME-TRAP very successfully boosts T-cell responses primed with a simian Adenovirus vector, inducing the highest level of CD4+ and CD8+ T-cell responses ever observed using a vectored vaccine and affording protection from malaria infection (A. Hill unpublished data).

For these reasons we now wish to assess an MVA construct encoding HCV NS that will be combined with AdCh3NSmut (or AdCh3NSmut1) in a heterologous prime/boost vaccination regimen to assess the safety and immunogenicity of this strategy in healthy and HCV infected patients. This study will address the following questions: In healthy volunteers:

1. Can vaccination with MVA-NSmut vector alone safely induce HCV specific T cell responses?
2. Can vaccination using a heterologous prime/boost vaccination schedule with AdCh3NSmut and MVA-NSmut safely induce HCV specific T cell responses?

   In HCV infected patients can a heterologous prime/boost vaccination schedule using AdCh3NSmut and MVA-NSmut:
3. Safely induce HCV specific T cell responses during pegylated-interferon and ribavirin (combination) therapy for HCV genotype-1 infection, after a significant decline in viral load, 14 weeks into therapy?
4. Safely induce HCV specific T cell responses during combination therapy for HCV genotype-1 infection, 2 weeks into therapy?
5. Safely induce HCV specific T cell responses in patients with chronic HCV (not receiving combination therapy) and a high viral load?
6. Suppress viral load in patients with chronic HCV, not on treatment with IFN and Ribavirin? Since the effect of combination therapy on HCV specific T cells is currently debated (see below) we will compare the T cell responses generated by the therapeutic prime/boost vaccination schedule in this study, to a group of matched historical control patients treated with combination therapy in whom immunological assessment has been made in an identical way to that proposed in this study.

ELIGIBILITY:
Inclusion Criteria:

The healthy volunteers must satisfy all the following inclusion criteria to be eligible for the study (group A1 or A2):

* Healthy adults aged 18 to 55 years (inclusive)
* Resident in or near the trial sites for the duration of the vaccination study
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* For women of child bearing potential, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination
* Men, including those with pregnant partners, should use barrier contraception until 3 months after the last vaccination
* Written informed consent

The patients with HCV in Groups B1, B2 and C1 must satisfy all the following inclusion criteria to be eligible for the study:

* HCV infected with genotype-1 infection (any viral load)
* Patients must not be currently receiving any treatment for HCV infection.
* Adults aged 18 to 64 years (inclusive)
* Resident in or near the trial sites for the duration of the vaccination study
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Liver transaminases may be within normal limits or elevated.
* For men in Arm B, including those with pregnant partners, a willingness to use barrier contraception until six months after completing treatment with IFN/ribavirin
* For women in Arm B, of child bearing potential, a willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination.
* For men in arm C, including those with pregnant partners, a willingness to use barrier contraception until three months after the last vaccination
* Written informed consent
* Patients with HCV in groups B1 and B2 must be treatment naïve to previous IFN and ribavirin combination therapy. They may be included if they have been previously treated with interferon monotherapy but relapsed after treatment.
* Patients with HCV in groups C1 may be treatment naïve, or have been previously treated with interferon monotherapy or interferon and ribavirin therapy and relapsed after treatment

Exclusion Criteria:

The subjects (both healthy individuals or patients) may not enter the study if any of the following exclusion criteria apply:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant simian or human adenoviral vaccine
* Clinical, biochemical (abnormal liver synthetic dysfunction defined by an elevated blood prothrombin time or a low blood albumin level), ultrasonographic, or liver biopsy (histology) evidence of cirrhosis or portal hypertension
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., Kathon
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Current suspected or known injecting drug abuse
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for HIV (antibodies to HIV) at screening
* Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or may influence the result of the study, or the patient's ability to participate in the study
* Any other finding which in the opinion of the investigators would significantly increase the risk of having an adverse outcome from participating in the protocol
* Individuals who have had a temperature >38°C in the 3 days preceding vaccination.
* Patients likely to have been infected with HCV within the last 12 months

In addition to the above listed exclusion criteria:

Patients with HCV may not enter arms B1 and B2 of the study if any of the following exclusion criteria applies:

* Patients are non-responders to previous IFN-alpha monotherapy
* Patients who received IFN-alpha and ribavirin or PEG-IFN and ribavirin in the past and who were non-responders or who relapsed during or after therapy
* Patients with a known allergy to ribavirin or interferon-alpha
* Haemoglobin less than 10g/dl
* Severe neutropenia or thrombocytopenia
* Patients who have had a heart attack or who have suffered from any other severe heart disease in the last 6 months
* Patients with haemoglobinopathies
* Autoimmune hepatitis
* Autoimmune disease
* History of organ transplantation
* Uncontrolled seizures
* Uncontrolled severe psychiatric conditions

Patients with HCV may not enter arm C if they were previous non-responders to interferon monotherapy, or interferon and ribavirin combination therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2010-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participant with adverse events, type and severity of adverse events | Different time frames depending on study groups
  To assess the safety of new hepatitis C vaccine candidates, AdCh3NSmut (and the improved version AdCh3NSmut1) and MVA-NSmut when administered to healthy volunteers and to HCV infected patients. The specific endpoints for safety will be actively collected data on adverse events.

SECONDARY OUTCOMES:
Immunogenicity | Different time frames depending on the study groups
  To assess the cellular immune response generated by AdCh3NSmut (and the improved version AdCh3NSmut1) and MVA-NSmut, when administered sequentially, to patients with hepatitis C virus infection. The specific endpoint of cellular immune response will be collected via IFN-gamma ELISpot assay and other exploratory immunological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Barnes, Dr., Study Chair — University of Oxford, UK; Paul Klenerman, Prof., Principal Investigator — University of Oxford, UK; David Gorard, Dr, Principal Investigator — Wycombe Hospital, High Wycombe, Buckinghamshire
Locations (3):
- United Kingdom (3):
  - Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire
  - John Radcliffe Hospital, Headley Way, Headington, Oxford
  - Wycombe Hospital, High Wycombe, Buckinghamshire, High Wycombe

REFERENCES:
- [Derived] Alsaleh G, Panse I, Swadling L, Zhang H, Richter FC, Meyer A, Lord J, Barnes E, Klenerman P, Green C, Simon AK. Autophagy in T cells from aged donors is maintained by spermidine and correlates with function and vaccine responses. Elife. 2020 Dec 15;9:e57950. doi: 10.7554/eLife.57950. PMID 33317695
- [Derived] Swadling L, Capone S, Antrobus RD, Brown A, Richardson R, Newell EW, Halliday J, Kelly C, Bowen D, Fergusson J, Kurioka A, Ammendola V, Del Sorbo M, Grazioli F, Esposito ML, Siani L, Traboni C, Hill A, Colloca S, Davis M, Nicosia A, Cortese R, Folgori A, Klenerman P, Barnes E. A human vaccine strategy based on chimpanzee adenoviral and MVA vectors that primes, boosts, and sustains functional HCV-specific T cell memory. Sci Transl Med. 2014 Nov 5;6(261):261ra153. doi: 10.1126/scitranslmed.3009185. PMID 25378645